CLINICAL TRIAL: NCT01337791
Title: Efficacy, Safety and Tolerability of Telbivudine in HBeAg Positive Chronic Hepatitis B Pregnant Women With Elevated Alanine Aminotransferase Levels
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Guo-Rong Han, The Second Affiliated Hospital of the Southeast University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H200804IRB
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Hepatitis B; Pregnancy Complications; High Viral Load; Elevated Alanine Aminotransferase Levels
Keywords: chronic hepatitis B; hepatitis B virus; perinatal transmission; Telbivudine
MeSH Terms: conditions — Hepatitis B, Chronic; Pregnancy Complications; Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (No Intervention)
  Interventions: Drug: Telbivudine treatment
- telbivudine (No Intervention)

INTERVENTIONS:
Drug: Telbivudine treatment — Two arms in this study, One is Telbivudine 600 mg by mouth daily from late pregnancy to 28 weeks of post partum. Another arm is clinical observation only without telbivudine treatment
  Arms: control

SUMMARY:
Telbivudine reduces DNA and normalizes alanine aminotransferase levels (ALT) in chronic hepatitis B patients with few adverse effects, but its use during pregnancy has not been explored. In this open-label, prospective study from the second trimester to post-partum week 28. This trial is to study the efficacy, safety and tolerability of Telbivudine in HBeAg Positive Chronic Hepatitis B Pregnant Women with high level of serum HBV DNA and elevated alanine aminotransferase levels.

ELIGIBILITY:
Inclusion Criteria:

* age between 20-40 years
* gestational age between 12-30 weeks
* serum HBsAg and HBeAg positivity
* HBV DNA levels >6log10 copies/mL
* ALT >1x ULN (40 IU/mL) and < 10x ULN.

Exclusion Criteria:

* co-infection with hepatitis A, C, D, E or HIV
* evidence of hepatocellular carcinoma; decompensated liver disease or significant renal, cardiovascular, respiratory or neurological co-morbidity
* concurrent treatment with immune-modulators, cytotoxic drugs, or steroids
* clinical signs of threatened miscarriage in early pregnancy
* evidence of fetal deformity by 3-dimensional ultrasound examination
* the biological father of the child had CHB

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The efficacy of Telbivudine treatment (DNA reduction, ALT normalization, and infants' immunoprophylaxis failure) and safety | From late pregnancy to 28 weeks of postpartum

SECONDARY OUTCOMES:
Changes in maternal HBeAg titers and lost/seroconversion of HBeAg or HBsAg | From late pregnancy to 28 weeks of postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gynecology and Obstetrics, The Second Affiliated Hospital of the Southeast University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Pan CQ, Han GR, Jiang HX, Zhao W, Cao MK, Wang CM, Yue X, Wang GJ. Telbivudine prevents vertical transmission from HBeAg-positive women with chronic hepatitis B. Clin Gastroenterol Hepatol. 2012 May;10(5):520-6. doi: 10.1016/j.cgh.2012.01.019. Epub 2012 Feb 14. PMID 22343511